CLINICAL TRIAL: NCT05736913
Title: Immunogenicity, Safety and Tolerability of Intradermal COVID-19 Vaccination Strategy in Immunocompromised Patients: a Prospective, Randomized Trial.
Brief Title: Intradermal COVID-19 Vaccination in the Immunocompromised
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW 21-214
Record Dates: First submitted 2023-02-19; First posted 2023-02-21 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: immunogenicity; safety; intradermal; COVID-19; vaccine; immunocompromised
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: prospective, open-labelled, randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradermal (Active Comparator): One dose of 30ug (0.3mL) intradermal BNT162b2
  Interventions: Biological: ID BNT162b2 vaccine
- Intramuscular (Active Comparator): One dose of 30ug (0.3mL) intramuscular BNT162b2
  Interventions: Biological: IM BNT162b2 vaccine

INTERVENTIONS:
Biological: ID BNT162b2 vaccine — intradermal BNT162b2 vaccine
  Arms: Intradermal
Biological: IM BNT162b2 vaccine — intramuscular BNT162b2 vaccine
  Arms: Intramuscular

SUMMARY:
COVID-19 is an infectious disease caused by SARS-CoV-2 virus, causing millions of deaths around the globe since the beginning of the pandemic. COVID-19 vaccination was proven to be effective at reducing both mortality and development of severe COVID-19 after infection. Vaccine-elicited protection is particularly important for immunocompromised patients, as they are more susceptible to infections with their defective immune response, for instance, previous review had suggested that patients with malignancies and recipients of solid organ transplants may be at increased risk of developing severe COVID-19 disease and even death.

To further complicate the scenario, there are two obstacles: firstly, immunocompromised individuals may have suboptimal response from vaccinations, as studies have shown that recipients of solid organ transplant have suboptimal or even are seronegative after the fourth dose booster vaccination . Secondly, with constant mutation of the SARS-CoV-2 viruses, new variants evolve over time, leading to reduction in vaccine efficacy and breakthrough infection in healthy individuals. Therefore, novel vaccine strategy should be considered to enhance the vaccine response in these immunocompromised individuals.

In this study, intradermal injection instead of intramuscular injection for vaccine delivery is proposed, as the investigators have observed improved immunogenicity and few adverse events from previous experience of influenza vaccination. The study aims to evaluate the immunogenicity, safety and tolerability of intradermal COVID-19 vaccination in immunocompromised patients.

DETAILED DESCRIPTION:
This is a randomized controlled trial performed in the Hong Kong West Cluster Hospitals under the Hospital Authority in Hong Kong. Immunocompromised individuals who completed two doses of COVID-19 vaccine are recruited and received a booster dose of BNT162b2 vaccine. Recruited individuals include patients who received solid organ transplant (SOT), patients who received stem cell or bone marrow transplant (SCBOT), patients who are undergoing chemotherapy or immunotherapy (COI) and patients who are receiving biologics therapy (BI). The study was approved by the institutional review board of the University of Hong Kong and Hospital Authority (UW 21-214).

After recruitment, participants are randomized to receive either one 30-μg dose (0.3 mL) of intramuscular BNT162b2 booster dose vaccination or one 30-μg dose (0.3 mL) of intradermal BNT162b2 booster dose vaccination. In addition, participants are further subdivided into different groups based on the priming vaccine received. Participant's blood samples are collected before booster vaccination (baseline), 28 days after booster dose, 3 months after booster dose and 6 months after booster dose vaccination. Blood samples collected are tested with live virus microneutralization assay (vMN), performed in the Biosafety level 3 facility of HKU to determine the level of neutralizing antibody in sera. Serial 2-fold dilutions of serum starting from 1:10 are incubated with 100 median tissue culture infectious doses (TCID50) of ancestral strain SARS-CoV-2, BA.1, BA.5.2, and XBB for 1.5 h at 37 °C. Then, a serum-virus mixture is added to VeroE6/TMPRSS2 cells (JCRB Cell Bank Catalogue no. JCRB1819) on 96-well plates. After 72 h of incubation at 37 °C and 5% CO2, the cytopathic effect (CPE) is examined and the antibody titre is determined by the highest dilution with 50% inhibition of CPE. In addition, A Surrogate SARS-CoV-2 neutralizing antibody (NAb) is performed to determine the level of NAb in serum sample. Testing is performed using a one-step competitive chemiluminescence immunoassay on the iFlash 1800 analyzer, as described in our previous study.

To assess the safety and adverse events of the vaccination, participants are asked to record any adverse events for 4 weeks after the booster dose.

The primary endpoint of this study is the vMN geometric mean titre (GMT) against WT, BA.1, BA.5.2 and XBB. The secondary endpoints are GMT fold increase and safety. Severe adverse events (SAEs) are defined as death, disabling or life-threatening conditions related to vaccine; Adverse events (AE) include fever (>38 °C), chills, headache, tiredness, nausea, vomit, diarrhea, muscle pain, joint pain, facial dropping, skin rash or injection site reactions (pain, redness, swelling, ecchymoses, itching).

ELIGIBILITY:
Inclusion Criteria:

1. Recruited subjects include adult subjects ≥18 years
2. Immunocompromised subjects as defined by the following.

   1. Patients who have undergone solid organ or stem cell transplantation and on immunosuppressive medication.
   2. Patients who are on chemotherapy, biologics or other immunosuppressive therapy.
   3. Patients who are on high-dose corticosteroid (prednisolone 0.5mg/kg daily or equivalent)
3. Negative IgG antibody response against Covid19 14 days after the second dose of Covid19 vaccination.
4. All subjects have to give written informed consent.
5. Subjects must be available to complete the study and comply with study procedures. Willingness to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response

Exclusion Criteria:

1. Inability to comprehend and to follow all required study procedures.
2. Have a recent history (documented, confirmed or suspected) of a flu-like disease within a week of vaccination.
3. Have a known allergy to polyethylene glycol (PEG) or other components of the study vaccines, or history of any anaphylaxis, serious vaccine reactions, to any excipients.
4. Have known active human immunodeficiency virus (HIV) infection.
5. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during this study. Unwilling to refuse participation in another clinical study through the end of this study.
6. Tympanic temperature ≥ 38°C within 3 days of intended study vaccination
7. Have a history of alcohol or drug abuse in the last 5 years.
8. Have any condition that the investigator believes may interfere with successful completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
vMN geometric mean titre | day 28 after vaccination
  microneutralization GMT

SECONDARY OUTCOMES:
vMN geometric meant titre fold increase | day 28 after vaccination
  microneutralization fold increase
Safety of the intradermal vaccination | day 28 after vaccination
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ivan FN Hung, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Anonymous patient's immunogenicity and safety data
Supporting Information: Study Protocol, CSR
Time Frame: 12 months
Access Criteria: email to the principal investigator

REFERENCES:
- [Result] Tawinprai K, Siripongboonsitti T, Porntharukchareon T, Wittayasak K, Thonwirak N, Soonklang K, Sornsamdang G, Auewarakul C, Mahanonda N. Immunogenicity and safety of an intradermal fractional third dose of ChAdOx1 nCoV-19/AZD1222 vaccine compared with those of a standard intramuscular third dose in volunteers who previously received two doses of CoronaVac: A randomized controlled trial. Vaccine. 2022 Mar 15;40(12):1761-1767. doi: 10.1016/j.vaccine.2022.02.019. Epub 2022 Feb 21. PMID 35210118
- [Result] Niyomnaitham S, Atakulreka S, Wongprompitak P, Copeland KK, Toh ZQ, Licciardi PV, Srisutthisamphan K, Jansarikit L, Chokephaibulkit K. Immunogenicity and reactogenicity of accelerated regimens of fractional intradermal COVID-19 vaccinations. Front Immunol. 2023 Jan 17;13:1080791. doi: 10.3389/fimmu.2022.1080791. eCollection 2022. PMID 36733395